CLINICAL TRIAL: NCT02328352
Title: The Buckypaper as a New Device in the Treatment of Some Solid Cancer and Hematopoietic System Tumors and as a New Fixing Device for Prosthetic Surgery. In Vivo Study on Effects of BP Implantation, Preliminary to Human Surgical Applications
Brief Title: "BP as a New Device for Surgery and Solid Cancer and Hematopoietic System Tumors Treatment. Effects of BP Implantation"
Acronym: DM159
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University of Sannio (Other); Appialab Veterinary Reseach Labaratory (Unknown); Catholic University of the Sacred Heart (Other); Istituto Superiore di Sanità (Other)
Responsible Party: Principal Investigator, Massimo Chiaretti, Dr, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DM SALUTE 159/2010 20/09/2010
Record Dates: First submitted 2014-06-24; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Hernia of Abdominal Wall; Incisional Hernia
Keywords: Buckypaper (BP) of Multi-Walled Carbon Nanotubes (MWCNTs); surgical hernia prosthesis; abdominal wall defects surgery; prosthesis adhesion; disaster preparation and recovery hernia; Abdominal Wall Disaster Surgery; Fixation of prosthetic materials in general surgery
MeSH Terms: conditions — Hernia, Abdominal; Incisional Hernia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BP selfstanding felt (Experimental): laparotomy intervention with the incision of 10 cm navel-pubis will be performed, splaying of the skin and subcutaneous layers, then will be incised the fascia plane, and muscles. Ten rabbits (hereafter defined as BPR1-BPR10) will receive 2x2cm2 samples of BP selfstanding felt in a pocket created between muscular fascia and large muscles of the abdominal wall.
  V-Loc 180 (ref VLOCL0024, lot. A1D0899)
  Interventions: Procedure: BP selfstanding felt
- PP mesh (Active Comparator): intervention of laparotomy with the incision of 10 cm navel-pubis will be performed, splaying of the skin and subcutaneous layers, then will be incised the fascia plane, and muscles. A 2x2cm2 sample of PP mesh was implanted without stitches into a pocket between large abdominal muscle and abdominal fascia.
  Other names: V-Loc 180 (ref VLOCL0024, lot. A1D0899) PR Parietene mesh Tyco (ref. PP3030, lot. SIK00587)
  Interventions: Procedure: PP mesh
- BP intraperitoneal mesh (Experimental): A surgical scar was performed on the abdominal linea alba and carried out deeply for entering into the abdominal cavity. In five rabbits (BPR21-BPR25). A 2x2cm2 BP intraperitoneal mesh was then be inserted with the rough side facing the parietal peritoneum surface and the smooth and brilliant surface facing to the visceral peritoneum and gut.
  Interventions: Procedure: BP intraperitoneal mesh
- control group (Active Comparator): Five rabbits (R26-R30) will be used as control group.
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: BP selfstanding felt — intervention of laparotomy with the incision of 10 cm navel-pubis will be performed, splaying of the skin and subcutaneous layers, then will be incised the fascia plane, and muscles. Ten rabbits (hereafter defined as BPR1-BPR10) will receive 2x2cm2 samples of BP selfstanding felt in a pocket created between muscular fascia and large muscles of the abdominal wall.
  Other Names: BP (Buckypaper NanoLab Inc., Newton, MA 02458 USA); V-Loc 180 (ref VLOCL0024, lot. A1D0899)
  Arms: BP selfstanding felt
Procedure: PP mesh — intervention of laparotomy with the incision of 10 cm navel-pubis will be performed, splaying of the skin and subcutaneous layers, then will be incised the fascia plane, and muscles. A 2x2cm2 sample of PR (polypropylene) prosthesis was implanted without stitches into a pocket between large abdominal muscle and abdominal fascia
  Other Names: Other names: V-Loc 180 (ref VLOCL0024, lot. A1D0899); PR Parietene mesh Tyco (ref. PP3030, lot. SIK00587)
  Arms: PP mesh
Procedure: BP intraperitoneal mesh — Laparotomy on the linea alba carried out deeply for entering into the abdominal cavity, a 2x2cm2 BP sample implantation with the rough side facing the parietal peritoneum surface and the smooth and brilliant surface facing to the visceral peritoneum and gut
  Other Names: BP (Buckypaper NanoLab Inc., Newton, MA 02458 USA); V-Loc 180 (ref VLOCL0024, lot. A1D0899)
  Arms: BP intraperitoneal mesh
Procedure: control group — observational intervention in 5 rabbits with the same body weight and the same age will be observed and will be feeded in the same way of the BP device intraperitoneal implanted group
  Other Names: famale 3000 gr New Zeeland rabbits (Harland)
  Arms: control group

SUMMARY:
Nanotechnologies applied to General Surgery and Emergency Surgery: The Buckypaper as a new fixing method for prosthetic materials in the treatment of abdominal wall hernias in humans, in laparotomic procedures and as a new device for the treatment of solid cancer and hematopoietic system tumors.

The experimentation on this new material, preliminary conducted on breed female rabbit New Zeeland, will be applicable to human, if the results in terms of toxicity and durability will be comfortable.

DETAILED DESCRIPTION:
The Buckypaper (BP) is an innovative material that has attracted the attention of many research groups engaged in the study of its possible applications in various technological fields preliminary to human experimentation. In fact the experimentation, preliminary conducted on animal model, will be applicable to human, if the results in terms of toxicity and durability will be comfortable.

The interesting material properties, such as good mechanical strength, electrical conductivity, low density, porosity adaptable, are closely associated to the intrinsic characteristics of carbon nanotubes (CNTs), of which BP is made . The high surface development of CNT, in addition to promoting their aggregation, allows the preparation of micro-and nano-porous membranes that exclude the passage of colloidal particles with a diameter greater than 50 nm. The microporous structure, also gives the BP high capacity to absorb liquids, such as water, for which the effect of capillarity, penetrates quickly in the mesh material . This could be a possible interpretation of the rapid and effective adhesion of BP to biological tissues observed in our studies on the effects of the material implanted in vivo. The bioadhesion of BP has been documented in ex vivo experiments mechanical peeling (bench surgery), conducted in advance using as substrate, guinea pig, rats, the abdominal muscle fascia of rabbits. The results showed that the force required the posting of BP from organic support is much greater than that required for the conventional prosthesis made from polymer networks, commonly used in hernia surgery fixed with glue and biological prosthetic material bioadhesive synthetic currently marketed . Based on these assessments and based on the potential offered by the use of BP in the field of prosthetic surgery, deductible by the intrinsic characteristics of the material in this project is expected to further research for the development of a new generation of prosthetic materials for use surgical -based BP, easily implantable by the surgeon without the need for sutures, graphs and / or biological glues . The reasons are:

1. stitches: they could tighten the knot vessels (ischemia-atrophy) or nerves (chronic pain);
2. graphs: placing blind and can cause bleeding or pain;
3. biological glues: derived from the plasma of donors and thus could transmit diseases unknown.

It is still unknown if BP has the appropriate mechanical properties to withstand the stresses that occur on the abdominal wall and In any case is documented the good bio-adhesion on living tissues and anatomical preparations, but only if made humid.

For this reason it was decided to prepare composite materials BP/polypropylene. Such materials, defined as "coupled", will be obtained by adhering on the smooth face of BP, a polymeric support which confers to the hybrid film, the correct mechanical resistance. Such a system may be subject to further changes. Indeed, exploiting the functional groups present or introduced into the crystalline structure of MWCNTs and/or on the polymer, it will be possible to implant on the muscle/muscular fascia surface, the composite material, to obtain gripping. Moreover, biologically active molecules, with functions antimicrobial, anti-adhesive, anti-inflammatory or analgesic, can be introduced into the crystalline structure of MWCNTs, for modulate the inflammatory response and the incorporation of the implanted material in the fibrous scar.

The objective of this project is to obtain results that can direct the search for the ultimate realization of a prosthetic device for use in abdominal surgery appliable to humans.

Our Research Group proposes that the present research program has all the skills to achieve all the objectives .

It brings together researchers with proven expertise and experience in various fields of General Surgery and Prosthetic Surgery of abdominal wall and Experienced scientist of Materials Science especially of polymeric nature, also for biomedical uses, Organic Chemistry, and synthesis of bio-conjugates for the development of slow release systems of drugs, characterization of biological systems through techniques of nuclear magnetic resonance (NMR). The surgeon in the unit of search, in fact, for many years been engaged both in the resolution of issues related to surgical techniques, both in the assessment of the effects on the living organism of conventional prosthetic materials and innovative ones, in the proposed project, including through in vivo testing, conducted according to a protocol specially prepared and approved by the Ministry of Health.

The protocol have been drawn in the respect of environmental policies, and ethical principles on experimentation on animal model, in accordance with the guidelines of the European Union (86/609/EEC-European Economic Community), and the Italian Law n° 116/92.

Will be conducted systematic experiments in 30 New Zealand female rabbits (R1-R30), weighting about 3000 g (Harlan Laboratories). The "in vivo" investigations will be about the biocompatibility and the adhesion of BP in the abdominal scar and in the performing of the intervention of incisional hernia and plastic surgery of the inguinal hernia.

The biocompatibility of the BP will be investigated by means of blood chemistry tests. Blood samples of 3 ml of whole blood will run to every beast after induction of general anaesthesia, from the ear vein, before surgery with prosthetic implant, and prior to euthanasia as indicated in the Time schedule.

Methodology and technique of the experiment :

These experiments are preliminar to human use and will be performed under general anesthesia with endotracheal intubation, then hair removal, disinfection and preparation of the surgical field. A midline incision of about 10 cm navel-pubis will be performed, splaying of the skin and subcutaneous layers, then will be incised the fascia plane, and muscles deep to enter in the peritoneum sac. The execution of the blood sampling coincident with the detection of the body weight and the execution of ultrasound of the abdominal region for the study of the implant site in search of signs of sepsis and incisional hernia.

We will implant this kind of new matherials on humans but before to this we will try to study the tollerability and toxicity on an animal model so drawn: ten rabbits (hereafter defined as BPR1-BPR10) (Buckypaper Rabbit subject 1 to 10) will receive 2x2cm2 samples of BP (Buckypaper) and ten rabbits will receive 2x2cm2 samples of PR (polypropylene) (PRR11-PRR20) in a pocket created between muscular fascia and large muscles of the abdominal wall. In five rabbits (BPR21-BPR25), the surgical incision will carried out on the abdominal linea alba and performed deeply, for entering into the abdominal cavity. The control group (R26-R30) will not undergo to surgery.

A 2x2cm2 BP sample will then be inserted with the rough side facing the parietal peritoneum surface and the smooth and brilliant surface facing to the visceral peritoneum (BPR21-BPR25). Five rabbits (R26-R30) will not be operated but will be used as control group. The animals will be monitored and controlled daily, during the entire studied period, in order to continually assess their state of health, and body weight. At the 35th day will be picked up a blood sample for examination. Finally the animals will be sacrificed under general anesthesia.

The cases BPR1-BPR10 (group A) will be compared with the PRR11-PRR20 (control group B) comparing the effects of implants of BP and the same size in Parietene already in use in reconstructive surgery of healthy man . After the intervention, that will last about 60 minutes from the time of induction, the animal will be slowly awakened and then brought back in the room housing.

At the time of sacrifice will be prepared anatomic samples of all the viscera and of the implantation site, to be studied histologically. Histopathological samples for microscopic examination will be prepared. Portions of BP implanted in BPR 1-BPR 10 will be excised with all the surrounding fascia, dermal and muscular tissues. The same procedures will be performed, also in PRR 11-PRR 20 group and BPR 21-BPR 25 group. The samples will be fixed in 10% buffered formalin, cut and stained with Haematoxylin and Eosin (H&E) for histological observation.

The post-operative pain, as in the human, it will be mild, and will be treated with analgesics according to techniques standardized in humans. In our experience, the animals undergo to prosthetic surgery, both the experimental and the control group, will treated with prophylactic antibiotics and pain medication in the immediate post -operative, and will be closely watched.

Even if in animal model, the sterility of all the surgical procedure prevents inflammation, edema and sepsis and abscesses and ensures a low level of postoperative pain. The days after the surgical procedure is expected a moderate appetite of the operated animals and mild clinical symptoms related to the post-operative .

All treated animals will be observed daily to carefully control the amount of food that will be consumed and thus the potential loss of appetite. Will be look for evidence of possible inflammatory and degenerative processes affecting the skin of the abdominal wall, the symptoms of infection or rejection of the prosthesis. If weight loss will be excessive (eg more than 10% of the normal weight of an animal of the same race, the same age and in comparison to the control group), or the animal will show clinical symptoms of suffering more than a normal postoperative, will be subjected to general anesthesia and then deleted.

The analgesic and antibiotic therapy performed in the postoperative period will be as follows :

Antibiotic : enrofloxacin 2.5 mg /kg /day I.M. for 5-7 days; and anti-inflammatory analgesic : ketoprofen, Findol 10%, 0.3 ml/10kg/die i.m. for 3-5 days. If necessary will be given also tramadol, 2-4 mg /kg/day in the first 2 /3 days post-intervention . The surgical wound will be checked daily.

The clinical-chemical parameters examined from blood samples of 3 ml will be: BUN (Blood Urea Nitrogen), blood glucose, creatinine, sodium, potassium, calcium, magnesium, albumin, total proteinemia and Blood protein level, SGOT(Serum Glutamic Oxaloacetic Transaminase), SGPT(Serum Glutamic PyruvateTransaminase), GGT(gamma glutamyl transferase), ALP(alkaline phosphatase) and fractionated bilirubin, PT(Prothrombin Time), APTT/PTT(Activated partial thromboplastin time), Fibrinogen, CBC(Complete Blood Count) formula, lymphocyte subpopulations, C-reactive protein, erythrocyte sedimentation rate.

Will be performed ultrasound examination to evaluate morphologically the prosthesis' incorporation, the formation of seroma, bruises, abscesses. This procedure will be performed under sedation and followed by body weight check and the pick-up of a blood sample. The same procedure will be repeated twice at the intervention and after 35 days at the sacrifice.

ELIGIBILITY:
Inclusion Criteria: animal model: New Zeeland female rabbits of 3000 gr of body weight -

Exclusion Criteria: any kind of illness in rabbit subjects

-

Ages: 3 Months to 6 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2010-10; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
number of moths without surgical hernia recurrence | 54 weeks
  Durability (in months) without recurrence of hernia and incisional hernia of surgical device.

SECONDARY OUTCOMES:
number of mm displacement from the point of implantation (at 12 weeks after BP implantation) | 3 months
  Ability (number of mm displacement from the point of implantation at 12 weeks after BP implantation) of the BP as bio-adhesive tape for prosthetic materials to avoid displacement of implanted prosthesis.
number of BP fragments in bioptic samples of Bowman capsule | 12 weeks
  toxicology of BP measured as number of BP fragments in bioptic samples of Bowman capsule of the nephron at 12 weeks
number of viable tumor cells in cultures after 48 hours of exposition to BP | 48 hours
  antineoplastic activity of BP device in the treatment of some solid cancer and hematopoietic system tumors: this item is measured ex vivo as the ability of BP to inhibit tumor cell replication (number of viable tumor cells in cultures after 48 hours of exposition to BP)

OTHER OUTCOMES:
delta of value of creatinine, transaminasis and PT, PTT, fibinogen from the T0 to 12 weeks. | 12 weeks
  toxicology of BP measured as modifications of values (delta) of creatinine, transaminasis and PT, PTT, fibinogen in blood samples from the T0 to 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Chiaretti, MD, PhD, MSc, Principal Investigator — University of Roma La Sapienza
Locations (1):
- National Health Institute (ISS Istituto Superiore di Sanità), Viale Regina Elena 299, Rome, Roma, Italy

REFERENCES:
- [Result] Martinelli A, Carru GA, D'Ilario L, Caprioli F, Chiaretti M, Crisante F, Francolini I, Piozzi A. Wet adhesion of buckypaper produced from oxidized multiwalled carbon nanotubes on soft animal tissue. ACS Appl Mater Interfaces. 2013 May 22;5(10):4340-9. doi: 10.1021/am400543s. Epub 2013 May 1. PMID 23635074
- [Result] Bellucci S, Chiaretti M, Onorato P, Rossella F, Grandi MS, Galinetto P, Sacco I, Micciulla F. Micro-Raman study of the role of sterilization on carbon nanotubes for biomedical applications. Nanomedicine (Lond). 2010 Feb;5(2):209-15. doi: 10.2217/nnm.09.100. PMID 20148633
- [Result] Bellucci S, Chiaretti M, Cucina A, Carru GA, Chiaretti AI. Multiwalled carbon nanotube buckypaper: toxicology and biological effects in vitro and in vivo. Nanomedicine (Lond). 2009 Jul;4(5):531-40. doi: 10.2217/nnm.09.36. PMID 19572819
- [Result] Di Sotto A, Chiaretti M, Carru GA, Bellucci S, Mazzanti G. Multi-walled carbon nanotubes: Lack of mutagenic activity in the bacterial reverse mutation assay. Toxicol Lett. 2009 Feb 10;184(3):192-7. doi: 10.1016/j.toxlet.2008.11.007. Epub 2008 Nov 21. PMID 19063954
- [Result] Catani M, De Milito R, Pietroletti R, Chiaretti M, Spaziani E, Leardi S, Simi M. Is there a place for intraperitoneal onlay mesh repair (IPOM) of inguinal hernia among laparoscopic techniques? Hepatogastroenterology. 2004 Sep-Oct;51(59):1387-92. PMID 15362760
- [Result] Catani M, De Milito R, Ratta G, Abati G, Chiaretti M, Rengo M. [Laparoscopy in an abdominal emergency: the diagnosis and therapy in 3 clinical cases of acute abdomen]. Ann Ital Chir. 1999 Mar-Apr;70(2):265-8; discussion 268-9. Italian. PMID 10434461
- See also: Carbon nanotubes toxicology and effects on metabolism and immunological modification in vitro and in vivo — http://iopscience.iop.org/0953-8984/20/47/474203/
- See also: prot. C26A10HCNR, founding of 35000€ Prof Lucio D'Ilario, Prof. Andrea Martinelli, Dott. Massimo Chiaretti , prot letter 0003306 project n° 304P25, interfaculty Chemistry Dep, General Surgery Paride Stefanini Dep. — http://www.uniroma1.it